CLINICAL TRIAL: NCT06873763
Title: A Single-arm, Phase Ib/2 Study of Nelmastobart in Combination With Trifluridine/Tipiracil and Bevacizumab in Metastatic/Recurrent Colorectal Cancer Patients With Resistance or Intolerance to Oxaliplatin and Irinotecan-based Chemotherapy
Brief Title: Nelmastobart in Combination With Trifluridine/ Tipiracil and Bevacizumab in Metastatic/ Recurrent Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: STCube, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STCUBE-003
Record Dates: First submitted 2025-02-17; First posted 2025-03-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer (CRC); Recurrent Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nelmastobart 800 mg+Trifluridine/Tipiracil+Bevacizumab (Experimental): 3 reducing doses of Trifluridine/Tipiracil will be administered to participants
  Interventions: Drug: Nelmastobart 800 mg+Trifluridine/Tipiracil+ Bevacizumab

INTERVENTIONS:
Drug: Nelmastobart 800 mg+Trifluridine/Tipiracil+ Bevacizumab — Trifluridine/tipiracil is dose-deescalated from 35 mg/m² to 30 mg/m² and 25 mg/m² to determine the RP2D, in combination with fixed doses of Nelmastobart and Bevacizumab, in patients with metastatic colorectal cancer who are refractory or intolerant to prior oxaliplatin- and irinotecan-based chemotherapy.

SUMMARY:
The objective of this multi-center, single-group, open-label Phase Ib/II study is to evaluate the safety, pharmacokinetics, and efficacy of nelmastobart in combination with trifluridine/tipiracil and bevacizumab in metastatic or recurrent colorectal cancer patients with resistance or intolerance to oxaliplatin- and irinotecan-based chemotherapy, and to determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), and the efficacy and safety of the combination therapy in BTN1A1-positive patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects who participate in the study must meet all of the following inclusion criteria.

1. Adults ≥19 years old at the time of written informed consent
2. Patients with histologically/cytologically confirmed metastatic/recurrent colorectal cancer after failure of, or not eligible for oxaliplatin and irinotecan-based standard anticancer therapy (If a subject had a radical surgery for colorectal cancer followed by adjuvant anticancer therapy, and the disease recurred during the adjuvant anticancer therapy or within 6 months from the end of the adjuvant anticancer therapy, the adjuvant anticancer therapy will be considered primary palliative therapy.)
3. Subjects with at least one evaluable lesion, or non-measurable but evaluable lesion according to RECIST v1.1
4. Subjects with ECOG performance status 0-1
5. Subjects with adequate bone marrow and body organ functions

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin count (Hgb) ≥ 9.0 g/dL
   * Platelet count ≥ 100 x 109/L
   * Serum creatinine ≤ ULN x 1.5 or serum creatinine clearance > 30mL/min
   * Total bilirubin ≤ 1.5 x ULN (Subjects with biliary obstruction may be enrolled if they meet the criterion after adequate biliary drainage.)
   * AST and ALT ≤ 3 x ULN in the absence of liver metastasis; or AST and ALT ≤ 5 x ULN in the presence of liver metastasis
6. Subjects with adequate cardiac function at the screening visit

   * QTc calculated using the Fredericia formula ≤ 480 msec (Those with QTc >480 msec may be enrolled if the mean of 3 consecutive QTc measurements is <480 msec.)
7. A negative serum β-HCG test within 14 days prior to IP dosing for women of childbearing potential
8. Subjects who agree, and are able to use during the study medically reliable methods of contraception as follows

   * To be eligible for enrollment, women of childbearing potential (all women who can have physiological pregnancy during IP treatment and for 6 months after the end of IP treatment unless they use appropriate methods of contraception) must use the following methods of contraception.
   * Subjects must refrain from any type of sexual intercourse, and persistent abstinence in daily life is recommended. Periodic abstinence (e.g., rhythm method, cervical mucus method, basal body temperature method, etc.) and withdrawal method are not acceptable methods of contraception.
   * Female sterilization procedures: Bilateral ovariectomy with or without hysterectomy; tubal ligation within 6 weeks prior to enrollment in this study. If the subject is confirmed to have childbearing potential based on the assessment of hormone level, only bilateral ovariectomy will be permitted.
   * Vasectomized partner (at least 6 months prior to screening). For women who participate in the study, the vasectomized partner must be the only partner during her participation in this study.
   * Men must use condoms during sexual intercourse during and after IP treatment (for 6 months after the last IP dose).
9. Life expectancy ≥3 months
10. Subjects who consent to sampling tumor tissues or collecting tumor tissue samples obtained within 2 years prior to the screening visit
11. Subjects who, after being fully informed of the study, voluntarily decide to participate in the study, provide written informed consent, and agree to comply with study procedures during the study

    [Inclusion criteria for the phase 2 study] Subjects who participate in the phase 2 study must meet all of the following criteria.
12. Subjects with Tumor Proportion Score (TPS) ≥50 based on immunohistochemistry (IHC) at the screening visit

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will be excluded from the study.

1. Patients who have hypersensitivity to the active ingredient of IP or any of its components (excipients)
2. Individuals who had cytotoxic chemotherapy within 14 days prior to randomization; treatment with IP in another clinical trial with the elapse of ≤2 weeks from the last dose of that IP or ≤5 folds the half-life of that IP; or treatment with monoclonal antibody therapy within the past 4 weeks
3. Uncontrolled serious infection
4. Confirmed PD during treatment with trifluridine/tipiracil for palliative care or confirmed recurrence within 6 months after the end of such treatment
5. Individuals requiring high-dose steroids (>10 mg/day prednisone or equivalent) or other immunosuppressants

   * However, these individuals may be enrolled in the following cases.
   * Short-term (<7 days) use of systemic corticosteroids that are considered standard of care will be allowed.
   * Subjects requiring intermittent use of bronchodilators, inhalant steroids, or local steroid injections will be allowed.
   * Replacement therapy (e.g., thyroxine, insulin, physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered as a type of systemic treatment and will be allowed.
6. Pregnant or lactating women
7. Individuals with a history of autoimmune disease requiring systemic treatment (i.e., use of disease modifying therapy, corticosteroids, or immunosuppressants) within 2 years prior to the screening visit (However, enrollment will be possible for subjects with vitiligo, psoriasis not requiring systemic treatment, type 1 diabetes mellitus, hypothyroidism stably managed with hormone replacement therapy, Sjogren's syndrome, or resolved pediatric asthma/atopy.)
8. Individuals with active central nervous system lesions (radiologically unstable or symptomatic brain lesions). With the exception of patients with meningeal metastasis, individuals who had radiotherapy or surgical treatment may be enrolled if there is evidence that the patient's condition is maintained without steroid therapy and that the disease of the brain lesion has not progressed for ≥4 weeks.
9. Individuals with a documented history of cerebrovascular events (stroke or transient ischemic attack), unstable angina pectoris, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class IV within 6 months prior to the screening visit
10. Patients with hypertensive encephalopathy or hypertension that is not adequately controlled with antihypertensives
11. Individuals with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonia; or with active pneumonia based on screening chest X-rays
12. Individuals who received allogeneic stem cell or solid organ transplants
13. Individuals who received live attenuated vaccines within 30 days prior to the screening visit. Examples of live vaccines include, but are not limited to measles, mumps, rubella, varicella/(varicella) zoster, yellow fever, rabies, bacillus Calmette-Guerin, and typhoid vaccines. Injectable seasonal influenza vaccines are generally killed virus vaccines and will be allowed. However, intranasal influenza vaccines are live attenuated vaccines and will not be allowed.
14. Individuals with a history of other primary cancers

    * However, enrollment will be possible for the following cancers.
    * Adequately treated skin cancer (basal cell or squamous carcinoma) that is not melanoma, superficial cervical cancer or stage 1 bladder cancer, completely resected thyroid cancer which did not metastasize and for which all treatment is completed (Scars must have been adequately treated prior to study enrollment).
    * Treated solid tumor with no evidence of recurrent disease at least 36 months prior to screening
15. Side effects of prior anticancer therapy that did not recover to Grade ≤1 (with the exception of alopecia)
16. Individuals who had radiotherapy in an extensive lesion involving ≥30 % of the bone marrow within 4 weeks prior to the screening visit or limited range radiotherapy for palliative care within 2 weeks
17. Patients who had major surgery within 4 weeks prior to the screening visit or who have not recovered from side effects of surgery
18. Patients who are unable to take drugs orally or who have a past history, or pathological findings of major gastrointestinal surgery that may affect the absorption of IP
19. Patients who have evidence of active infection including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV)

    * However, enrollment will be possible for the following cases.
    * Patients with positive hepatitis B surface antigen (HBsAg) may be enrolled if HBV DNA is negative based on a local test.
    * Patients with positive hepatitis B core antibody (IgG anti-HBc) and a history of HBV infection may be enrolled if HBV DNA is negative.
    * Patients with positive anti-HCV Ab may be enrolled if HCV RNA is negative.
20. Patients with hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
21. Individuals with medical, psychiatric, or cognitive disorders or impaired ability to understand information, provide prior consent, comply with protocol procedures, or complete the study
22. Those whom the investigator deems inappropriate for participation in this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | up to 6 months
  Status of DLT will be presented with frequency, percentage and its 95% confidence interval (CI).
RP2D(Recommended Phase 2 Dose) | up to 2 years
  The recommended phase 2 dose (RP2D) of nelmastobart in combination with trifluridine/tipiracil and bevacizumab
MTD(Maximum Tolerated Dose) | up to 2 years
  To find the maximum tolerated dose (MTD)
Progression Free Survival (PFS) rate | up to 2 years
  Time from the start of treatment to objective tumor progression or all-cause death will be presented with survival curve, median survival time and its 95% CI using the Kaplan-Meier estimation.

SECONDARY OUTCOMES:
Phase 2 study; Overall Survival (OS) | up to 2 years
  Time from the start of treatment to all cause death
Phase 2 study; Objective Response Rate (ORR) | up to 2 years
  Investigator assessed ORR defined by RECIST 1.1 or iRECIST
Maximum plasma concentration (Cmax) | up to 6 months
  Maximum plasma concentration of Nelmastobart to evaluate PK parameters
Phase 2 study; Disease Control Rate (DCR) | up to 2 years
  Investigator assessed DCR at 16 weeks defined by RECIST 1.1 or iRECIST
PFS(Progression free survival) | up to 2 years
  Time from first dose until the date of objective disease progression or death
Phase 2 study; Duration of Response (DOR) | up to 2 years
  Time from the date of first confirmed objective response (CR or PR) after investigational drug administration to the first documented disease progression (PD) or death from any cause, with documentation of disease progression status and cause of death
AEs(Adverse Events) | up to 2 years
  Status of AEs will be presented with frequency, percentage and its 95% CI. AEs will be classified by SOC and PT of MedDRA (latest version) and presented with frequency, percentage and its 95% CI.
Tmax(Time to Maximum Plasma Concentration) | up to 2 years
  Time to reach Tmax of Nelmastobart to evaluate the PK parameters.

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, KR
  - Severance Hospital, Seoul, KR
  - Asan Medical Center, Seoul, KR
  - Korea University Anam Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No